CLINICAL TRIAL: NCT02263651
Title: Dead Space Closure With Quilting Suture Versus Conventional Closure With Drainage in Prevention of Seroma Formation After Mastectomy for Breast Cancer : a Randomized Controlled Trial
Brief Title: Dead Space Closure With Quilting Suture Versus Conventional Closure With Drainage
Acronym: QUISERMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PHRCK13 - LO / QUISERMAS; 2014-A00901-46 (Other: ID RCB); 140730B-12 (Other: ANSM)
Record Dates: First submitted 2014-09-29; First posted 2014-10-13 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Mastectomy; Seroma; Quilting suture
MeSH Terms: conditions — Breast Neoplasms; Seroma | interventions — Drainage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closure with conventional technique with drainage (Active Comparator): The skin flaps are not fixed subcutaneously but sutured at the edges, a closed suction drain is inserted under the flaps in the dead space created by the dissection at the pectoral area. The drain is stitched to the skin.
  Interventions: Procedure: Conventional closure with drainage
- Quilting suture without drainage (Experimental): In an attempt to obliterate the dead space, the skin flaps are sutured to the underlying pectoralis major with multiple parallel rows of 0/0 vicryl (or equivalent). Running sutures at periodic intervals (<2cm) are placed from the skin flaps to the underlying muscle.
  Interventions: Procedure: Quilting suture without drainage

INTERVENTIONS:
Procedure: Quilting suture without drainage — In an attempt to obliterate the dead space, the skin flaps are sutured to the underlying pectoralis major with multiple parallel rows of 0/0 vicryl (or equivalent). Running sutures at periodic intervals (<2cm) are placed from the skin flaps to the underlying muscle. Minor dimpling is considered acceptable and is expected to resolve. If severe dimpling is observed, stitches are removed and replaced.
  Efficiency of quilting suture relies on a rigorous repartition of the sutures with a special attention taken to the obliteration of the largest potential dead spaces and the empty axillary apex.
  The skin edges are sutured as stated before for the control group. Closed suction will not be used for draining the pectoral area.
  Other Names: Quilting suture
  Arms: Quilting suture without drainage
Procedure: Conventional closure with drainage — The skin flaps are not fixed subcutaneously but sutured at the edges, a closed suction drain is inserted under the flaps in the dead space created by the dissection at the pectoral area. The drain is stitched to the skin.
  The skin is closed in two layers with absorbable sutures, a deep layer of 2.0 or 3.0 vicryl sutures or equivalent, and a subcuticular closure with absorbable 3.0 or 4.0 Monocryl sutures or equivalent.
  Other Names: Conventional closure
  Arms: Closure with conventional technique with drainage

SUMMARY:
The objective of this study is to compare quilting suture of the "dead space" without drainage of the pectoral area to conventional closure with drainage to prevent post-operative seroma requiring intervention (aspiration or surgical intervention) within 21 days after mastectomy for breast cancer.

DETAILED DESCRIPTION:
Eligible patients are patients with operable breast cancer (invasive carcinoma and/or carcinoma in situ) for whom mastectomy is recommended or preferred by the patient either alone or in association with sentinel lymph node biopsy or standard level I/II axillary node dissection

Randomization will be stratified by center and by type of surgery (mastectomy alone/ mastectomy with sentinel node biopsy / mastectomy with axillary lymph node dissection).

Two follow-up visits will be performed: at 21 days and 9 months after surgery, these appointments are conventional, thus our trial will not modify usual follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years and ≤ 85 years
* Women with operable breast cancer (invasive carcinoma and/or carcinoma in situ) for whom mastectomy is recommended or preferred by the patient either alone or in association with sentinel lymph node biopsy or standard level I/II axillary node dissection
* Women that give her informed written consent
* French social security affiliation

Exclusion Criteria:

* Any physical or psychiatric condition that could impair with patient's ability to cooperate with postoperative data collection.
* Women with indication of bilateral mastectomy or immediate reconstruction.
* Degenerative neuromuscular disease with thoracic muscular damage
* Planned ambulatory surgery

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2014-10; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Wound seroma requiring aspiration or surgical intervention | Within 21 days following mastectomy
  A seroma is defined as a postoperative fluid collection via palpation on clinical examination. The Common Terminology Criteria for Adverse Events (CTCAE) which is a descriptive terminology that can be used for adverse event reporting provide a grading scale for seromas (lymphoceles).
  Only grade 2 and 3 seromas i.e. seromas requiring one or more aspirations or a surgical intervention will be considered as primary outcome.

SECONDARY OUTCOMES:
Wound seroma requiring aspiration or surgical intervention | Within 9 months following mastectomy
Wound seroma whatever their type (requiring or not intervention) | Within 21 days following mastectomy
Wound seroma whatever their type (requiring or not intervention) | Within 9 months following mastectomy
Other wound complications | Within 21 days following mastectomy
Other wound complications | Within 9 months following mastectomy
Surgical morbidity | During surgical intervention
Pain | Before surgery, day 1, 21 days and 9 months following mastectomy
  Visual Analogue Scale
Homolateral shoulder movement | Before surgery, 21 days and 9 months following mastectomy
  The range of arm movement scored from 1 to 4 according to estimated angles of arm abduction as 1 (less than 90°), 2 (90-134°), 3 (135-179°) and 4 (180°)
Cosmesis results | 21 days, 9 months following mastectomy
  Cosmetic results will be documented by patient,surgeon and by an blinded adjudication committee with possible response = poor, acceptable, good and excellent
Health related quality of life : EQ-5D-5L | Before surgery, day 1, 21 days and 9 months following mastectomy
  The descriptive system comprises 5 dimensions : mobility, self care, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems
Cost-effectiveness assessment | During the whole follow-up period i.e. 9 months following mastectomy
  Incremental net monetary benefice

CONTACTS AND LOCATIONS:
Overall Officials: Lobna OULDAMER, MD, Principal Investigator — University Hospital, Tours
Locations (6):
- France (6):
  - Conception Hospital, Marseille
  - Institut POALI-CALMETTES, Marseille
  - Institut de Cancérologie de l'Ouest, Nantes
  - CHU de Poitiers, Poitiers
  - Alliance Clinic, Saint-Cyr-sur-Loire
  - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ouldamer L, Bonastre J, Brunet-Houdard S, Body G, Giraudeau B, Caille A. Dead space closure with quilting suture versus conventional closure with drainage for the prevention of seroma after mastectomy for breast cancer (QUISERMAS): protocol for a multicentre randomised controlled trial. BMJ Open. 2016 Apr 4;6(4):e009903. doi: 10.1136/bmjopen-2015-009903. PMID 27044574